CLINICAL TRIAL: NCT03546244
Title: Effects of Musical Treadmill Training vs Traditional Treadmill Training on Gait Parameters in Patinets With Parkinson's Disease
Brief Title: Evaluation of Efficacy of Musical Treadmill in PD Rehabilitation
Acronym: EMTPDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Luca Sebastianelli, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Musical Treadmill in PD
Record Dates: First submitted 2018-05-08; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic; Treadmill
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- musical treadmill (Experimental): 4-week daily musical treadmill training, consisting in two session, 20 minute per session
  Interventions: Behavioral: musical treadmill
- traditional session (Active Comparator): 4-week daily traditional treadmill training, consisting in two session, 20 minute per session
  Interventions: Behavioral: Traditional treadmill

INTERVENTIONS:
Behavioral: musical treadmill — Patients will undergo a 4-week, 2 daily, incremental session of training with musical treadmill
  Arms: musical treadmill
Behavioral: Traditional treadmill — Patients will undergo a 4-week, 2 daily, incremental session of training with traditional treadmill
  Arms: traditional session

SUMMARY:
In order to evaluate the effectiveness of musical treadimll on gait parameters in patients with Parkinson's Disease, the investigators compare the outcome measures on two group of patients: one will undergo a 4-week daily musical treadmill training and one will undergo a 4-week daily traditional treadmill training

DETAILED DESCRIPTION:
Gait is altered in Parkinson's disease (PD) patients. It has been shown that treadmill training is useful in improving the gait's parameters in patients in early-moderate stages of disease. Moreover, it has been shown that the music, exploiting the entrainment, is effective in order to ameliorate several gait parameters, as step lenghts and cadence. No data are available about the effectiveness of the association between treadmill and music. The aim of this study is to evaluate the effect of a gait training using musical treadmill in patients in stages I-II-III Hoehn & Yahr (H&Y).

100 patients with PD in early-moderate stage of disease will be enrolled. All patients will undergo an intensive treatment: 2 session of 20-minutes treadmill training per day, 5 times a week, for 4 weeks. Treadmill speed will be previously set at 20% less the confidence speed and progressively increased of 20%. All patients will be evaluat at the enrolment and at the end of the treatment. The outcome misures are: 6 Minute Walking Test and Timed Up and Go Test.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2.5-3 according to the Hoehn and Yahr scale (H&Y);
* Stable pharmacological treatment for the last 6 weeks before the enrolment and during the hospitalization;
* Mini Mental State Examination (MMSE) ≥ 24;

Exclusion Criteria:

* Any focal brain lesion detected in brain imaging studies (CT or MRI) performed in the previous 12 months;
* Drug-induced dyskinesias;
* Disturbing resting and/or action tremor, corresponding to scores 2-4 in the specific items of UPDRS III;
* Behavioral disturbances (evaluated with Neuropsychiatric Inventory);
* Visual and auditory dysfunctions according to the general clinical evaluation and medical history;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2019-01-03 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Walking Test | 4 week
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes
Timed up and Go Test | 4 week
  The TUG is aimed to measure the ability of patients to perform sequential locomotor tasks that incorporate walking and turning

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's disease, Movement Disorders and Brain Injury Rehabilitation, "Moriggia-Pelascini" Hospital - Via Pelascini, 3, 22015, Gravedona ed Uniti, Como, Italy
Locations (1):
- Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No